CLINICAL TRIAL: NCT03313063
Title: Myocardial Characterization With Magnetic Resonance Imaging in Patients After Preeclampsia (Pilot Study)
Brief Title: Post-Pregnancy Cardio Trial
Acronym: PPC1
Status: Completed | Type: Observational
Sponsor: Charite University, Berlin, Germany (Other)
Responsible Party: Principal Investigator, Florian Herse, PhD, Charite University, Berlin, Germany
Other Study IDs: PPC1
Record Dates: First submitted 2017-10-13; First posted 2017-10-18 (Actual); Last update posted 2018-07-26 (Actual); Status verified 2018-07

CONDITIONS: Preeclampsia
Keywords: magnetic resonance imaging; myocard; preeclampsia
MeSH Terms: conditions — Pre-Eclampsia

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- PE: Women with a history or preeclampsia, between 18 - 50 years of age, 0.5 - 20 years postpartum
- Control: Age-matched women without any birth complications, between 18 - 50 years of age, 0.5 - 20 years postpartum

SUMMARY:
Preeclampsia is a systemic pregnancy disorder and is associated with an increased cardiovascular risk later in life. This study will characterize myocardial tissue in patients after preeclampsia compared to controls and investigate potential functional and structural changes in the heart of preeclamptic women primarily with two methods: cardiovascular magnetic resonance imaging and echocardiography. A comparison between these two methods, where appropriate, is also envisaged.

ELIGIBILITY:
Inclusion Criteria:

* postpartal window: 0.5 - 20 years
* cases: diagnosis of preeclampsia during the index pregnancy
* controls: age and BMI matched

Exclusion Criteria:

* metal implants
* kidney insufficiency (GFR < 30 ml/min/)
* claustrophobia
* contrast medium allergy
* current pregnancy/ lactation
* chronic hypertension (> 140/90)
* diagnosis of previous cardiovascular disease
* body weight over 120 kg
* big tattoos in thorax area

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Women between 18 and 50 years of age, 0.5 - 20 years postpartum either with preeclampsia diagnosis during index pregnancy or without pathological findings. Controls are matched to cases based on age and BMI.
Sampling Method: Non-Probability Sample
Enrollment: 47 (Actual)
Dates: Start 2017-08-28 (Actual); Primary Completion 2018-06-30 (Actual); Study Completion 2018-06-30 (Actual)

PRIMARY OUTCOMES:
any structural or functional change of the heart (combined outcome) | 0.5 - 20 years after delivery
  Combined outcome: myocardial fibrosis, edema, fat infiltrates, inflammation, reduced ejection fraction, hypertrophy

SECONDARY OUTCOMES:
myocardial fibrosis | 0.5 - 20 years after delivery
myocardial edema | 0.5 - 20 years after delivery
myocardial fat infiltrates | 0.5 - 20 years after delivery
myocardial inflammation | 0.5 - 20 years after delivery
myocardial hypertrophy | 0.5 - 20 years after delivery
reduced ejection fraction | 0.5 - 20 years after delivery

CONTACTS AND LOCATIONS:
Locations (1):
- Experimental and Clinical Research Center (ECRC), Berlin, Germany